CLINICAL TRIAL: NCT02535546
Title: Characterisation of Isolates of Streptococcus Pneumoniae in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Seasonal Trends in Pneumococcal Carriage in COPD Patients
Acronym: Helios
Status: Completed | Type: Observational
Sponsor: Beaumont Hospital (Other)
Responsible Party: Principal Investigator, Professor Richard Costello, Professor Richard Costello, Beaumont Hospital
Other Study IDs: BeamontH
Record Dates: First submitted 2015-08-26; First posted 2015-08-28 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic obstructive pulmonary disease (COPD); Streptococcus pneumoniae; Pneumonia; Pneumococcal conjugate vaccine-13 (PCV-13); Pneumococcal polysaccharide vaccine-23 (PPV-23); Pneumococcal vaccine
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputum
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients suffering from chronic obstructive pulmonary disease (COPD) commonly get exacerbations of their illness which have many potential triggers including infection. The most common cause of lung infection/pneumonia is an organism named Streptococcus pneumoniae. In Ireland a 13-valent pneumococcal conjugated vaccine (PCV-13) was recently introduced into the childhood vaccination programme. This study aims to investigate the carriage rate of S. pneumoniae in COPD patients over one year and to determine if isolates of S. pneumoniae found within the COPD population would be covered by the PCV-13 vaccine.

DETAILED DESCRIPTION:
This study aims to determine the potential contribution of S. pneumoniae to the morbidity of patients with COPD in Ireland and if the PCV-13 has potential for reducing infective exacerbations in this cohort. A group of 150 COPD patients are being monitored at quarterly intervals over one year. At each study visit patients report changes to COPD-related medication, recent hospitalisations and exacerbations and provide a sputum sample (or pharyngeal swab if not possible) which is assessed for the presence of S. pneumoniae.

The specific objectives of the study are:

1. To monitor the carriage rate of pneumococci in a cohort of Irish patients with COPD during and outside periods of acute exacerbation over a one year period.
2. To assess the COPD exacerbation rate amongst this group of patients.
3. To monitor changes in the proportion of patients positive for pneumococci carriage over a full season and to document those patients intermittently or permanently colonised.
4. To characterise S. pneumoniae isolates carried by COPD patients in terms of their genetic evolution, comparison with strains in other countries, and antimicrobial susceptibility.
5. To assess the proportion of colonised COPD patients that would be covered by current and future pneumococcal vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age.
* Have a clinical diagnosis of COPD.
* Have a forced expiratory volume at one second/forced vital capacity (FEV1/FVC) ratio < 80%.

Exclusion Criteria:

* Patients too unwell.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A combination of COPD inpatients and outpatients from Beaumont Hospital, Dublin, Ireland.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Carriage rate of Streptococcus pneumoniae in patients with COPD over four seasons. | One year.
  Patients with COPD are being monitored over a one year period for carriage of S. pneumoniae. Carriage is determined by analysis of sputum or pharyngeal swab samples which are collected from patients at quarterly intervals.

SECONDARY OUTCOMES:
Characterisation of carriage isolates of Streptococcus pneumoniae from COPD patients. | One year.
  Any carriage isolates of S. pneumoniae isolated from COPD patients are assessed for serotype and antibiotic resistance profiles to determine if they are covered by current pneumococcal vaccines.

OTHER OUTCOMES:
Correlation between seasonality and disease severity in COPD patients. | One year.
  COPD patients are met with at quarterly intervals over one year. At each meeting patients report recent COPD exacerbations, hospitalisations and medication use, as well as scores for disease severity. This data is being used to determine if there is a correlation between disease severity and the seasons in COPD patients.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Costello, Principal Investigator — Professor of Respiratory Medicine
Locations (1):
- RCSI Education and Research Centre, Beaumont Hospital, Dublin, Ireland

REFERENCES:
- [Background] Vickers I, O'Flanagan D, Cafferkey M, Humphreys H. Multiplex PCR to determine Streptococcus pneumoniae serotypes causing otitis media in the Republic of Ireland with further characterisation of antimicrobial susceptibilities and genotypes. Eur J Clin Microbiol Infect Dis. 2011 Mar;30(3):447-53. doi: 10.1007/s10096-010-1108-7. Epub 2010 Nov 13. PMID 21076929
- [Background] Vickers I, Fitzgerald M, Murchan S, Cotter S, O'Flanagan D, Cafferkey M, Humphreys H. Serotype distribution of Streptococcus pneumoniae causing invasive disease in the Republic of Ireland. Epidemiol Infect. 2011 May;139(5):783-90. doi: 10.1017/S0950268810001743. Epub 2010 Jul 19. PMID 20642870
- [Derived] McCarthy H, Jackson M, Corcoran M, McElligott M, MacHale E, Sulaiman I, Cushen B, Costello RW, Humpreys H. Colonisation of Irish patients with chronic obstructive pulmonary disease by Streptococcus pneumoniae and analysis of the pneumococcal vaccine coverage: a non-interventional, observational, prospective cohort study. BMJ Open. 2017 Jul 9;7(7):e013944. doi: 10.1136/bmjopen-2016-013944. PMID 28694340